CLINICAL TRIAL: NCT01425502
Title: Data-driven Quality Improvement in Primary Care: Cluster Randomised Controlled Trial to Test the Effectiveness of a Multifaceted Intervention in Reducing High Risk Prescribing of Non-steroidal Anti-inflammatory Drugs and Antiplatelet Agents
Brief Title: Data-driven Quality Improvement in Primary Care - Trial
Acronym: DQIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Dundee (Other)
Collaborators: NHS Tayside (Other Government); NHS Fife (Other Government)
Responsible Party: Principal Investigator, Bruce Guthrie, Professor of Primary Care Medicine, University of Dundee
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2011PS05; ARPG/07/2 (Other Grant/Funding Number: Chief Scientist Office)
Record Dates: First submitted 2011-08-26; First posted 2011-08-30 (Estimated); Last update posted 2016-02-02 (Estimated); Status verified 2016-01

CONDITIONS: Drug Safety
Keywords: High risk prescribing; Primary care; Non-steroidal anti-inflammatory drugs; Anti-platelet agents; Stepped wedge design; Cluster randomised controlled trial; United Kingdom

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- All practices (Other): The design is a stepped-wedge cluster randomised trial. All participating practices therefore receive the intervention at a start time which is randomised.
  Interventions: Behavioral: DQIP Intervention

INTERVENTIONS:
Behavioral: DQIP Intervention — The DQIP intervention comprises of:
  * Educational outreach
  * Information technology application
  * Financial incentives

SUMMARY:
A cluster randomised controlled trial to test the effectiveness of an informatics tool, educational and financial incentives to reduce high risk prescribing of non-steroidal anti-inflammatory drugs and anti-platelet agents.

DETAILED DESCRIPTION:
The trial described here is part of a programme which aimed to design a complex, primary care prescribing safety improvement intervention and test its effectiveness in a randomised controlled trial.

Non-steroidal anti-inflammatory drugs (NSAIDs) and antiplatelet drugs such as low dose aspirin and clopidogrel are responsible for a significant proportion of hospital admissions due to preventable adverse drug events (ADE), and are the drugs most commonly associated with fatal ADEs. Previous research has identified groups of patients and patterns of co-prescription in which use of these drugs is particularly high-risk , and national prescribing and safety guidance has embedded this research in clear recommendations to either avoid prescribing or to do so only when there is no alternative, and with caution. In previous epidemiological work, we have shown that high-risk use of NSAIDs, aspirin and clopidogrel is common, and pilot work in four practices has shown that focused review of prescribing by the practice reduced the targeted high-risk NSAID prescribing by approximately 40% after one round of feedback. This effect size is consistent with the PINCER trial where the intervention was a pharmacist facilitated review process.

We hypothesise that a multi-faceted intervention comprising of (1) educational outreach, (2) use of an informatics tool to monitor prescribing patterns at practice level and to prompt and facilitate the review of individual patients at risk of ADEs and (3) a small financial incentive to review patients will reduce rates of high-risk prescribing.

The specific research questions addressed by the trial are:

1. Does the intervention reduce the specified primary outcome of a composite measure of high risk non-steroidal anti-inflammatory drug, aspirin and clopidogrel prescribing?
2. Does the intervention reduce the specified secondary outcomes of: the nine individual measures constituting the composite; related admissions to hospital; repeat vs new prescribing?
3. If found to be effective, then is the intervention cost-effective?

The trial will use a stepped-wedge design, which is particularly suited to a sequential roll-out of an intensive and informatics based intervention focusing on patient safety. In this design, all participating practices receive the intervention, but are randomised to a starting time. At the point of entering the intervention phase of the trial, all practices will receive an educational outreach visit which will include training in the use of the informatics tool.

The informatics tool will provide regular feedback of any change in rates of high-risk prescribing for each individual measure and the composite measure, with the ability to drill-down to individual patient level and review a summary of each patient's relevant conditions and prescribing.

ELIGIBILITY:
Inclusion Criteria:

* General medical practices in NHS Fife and NHS Tayside with a compatible clinical IT system and agreeing to participate.
* Practices that agree to have relevant medication related data to be automatically extracted from their electronic clinical information systems from 1/10/10 to 30/9/13 (ie 12 months before first practice starts till 12 months after last practice starts).

Exclusion Criteria:

* Practices that use General Practice Administration System for Scotland (GPASS) or Egton Medicine Information System (EMIS) on the date of randomisation, since data extraction for the informatics requires Vision practice IT system.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2012-09; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Composite: Proportion of patients with any risk factor as defined in secondary outcome measures to 9, who have received any high risk prescriptions of anti-inflammatory drugs or antiplatelets as defined in secondary outcome measures 1 to 9 | 8 weeks
  The primary and all secondary outcome measures will be measured in each practice at 8 weekly intervals (reflecting that all measures assess high risk prescriptions for NSAIDs and antiplatelets in the last 8 weeks). At the time of initial data extraction, 8 weekly intervals will be constructed for the 12 months before the intervention start date.

SECONDARY OUTCOMES:
1. Proportion of patients with a history of peptic ulcer (risk factor), who have been prescribed a traditional* oral non-steroidal anti-inflammatory drug (NSAID) without gastro-protection (high risk prescription) | 8 weeks
  * a 'traditional' NSAID refers to any agent within this class except Cox 2 selective agents ('coxibs')
2. Proportion of patients aged 75 or over (risk factor), who have been prescribed a traditional* NSAID without gastro-protection (high risk prescription) | 8 weeks
3. Proportion of patients aged 65 or over and prescribed low dose aspirin (risk factor), who have been prescribed a traditional oral NSAID without gastro-protection (high risk prescription) | 8 weeks
4. Proportion of patients aged 65 or over and prescribed low dose aspirin (risk factor), who have been co-prescribed clopidogrel without gastro-protection (high risk prescription) | 8 weeks
5. Proportion of patients prescribed warfarin (risk factor), who have been co-prescribed a traditional NSAID without gastro-protection (high risk prescription) | 8 weeks
6. Proportion of patients prescribed warfarin (risk factor), who have been co-prescribed low dose aspirin or clopidogrel without gastro-protection (high risk prescription) | 8 weeks
7. Proportion of patients with a documented diagnosis of heart failure (risk factor), who have been prescribed an analgesic dose NSAID (high risk prescription) | 8 weeks
8. Proportion of patients prescribed both a diuretic and an ACE inhibitor/ Angiotensin Receptor Blocker (risk factor), who have been prescribed an analgesic dose NSAID (high risk prescription) | 8 weeks
9. Proportion of patients with a documented diagnosis of chronic kidney disease stage 3,4 or 5, who have been prescribed an analgesic dose NSAID (high risk prescription) | 8 weeks
10. Proportion of patients with any risk factor listed in secondary outcomes measures 1 to 6, who have been prescribed any high risk prescription listed in secondary outcome measures 1 to 6 | 8 weeks
11. Proportion of patients with any risk factor listed in secondary outcome measures 8 to 9, who have been prescribed any high risk prescription listed in secondary outcome measures 8 to 9 | 8 weeks
12. No. of patients admitted to hospital for gastro-intestinal bleeding AND high risk prescription as defined in secondary outcome measure 10, divided by patient months with gastro-intestinal risk factors as defined in secondary outcome measure 10 | 48 weeks
13. No. of patients admitted to hospital for heart failure exacerbation AND high risk prescription as defined in secondary outcome measure 7, divided by patient months with documented heart failure as defined in secondary outcome measure 7 | 48 weeks
14. No. of patients admitted to hospital for acute renal failure, dehydration or diarrhoea AND high risk prescription as defined in secondary outcome measure 11, divided by patient months with renal risk factors as defined in outcome measure 11 | 48 weeks
15. No. of patients admitted to hospital for gastro-intestinal bleeding, divided by patient months with gastro-intestinal risk factors as defined in secondary outcome measure 10 | 48 weeks
16. No. of patients admitted to hospital for heart failure exacerbation, divided by patient months with documented heart failure as defined in secondary outcome measure 7 | 48 weeks
17. No. of patients admitted to hospital for acute renal failure or with dehydration or diarrhoea (both defined as potentially inappropriate/ambulatory care sensitive admissions), divided by patient months with renal risk factors as defined in measure 11 | 48 weeks
18. No. of patients with any emergency admission to hospital, divided by patient months with gastro-intestinal risk factors as defined in secondary outcome measure 10 | 48 weeks
19. No. of patients with any emergency admission to hospital, divided by patient months with documented heart failure as defined in secondary outcome measure 7 | 48 weeks
20. No. of patients with any emergency admission to hospital, divided by patient months with renal risk factors as defined in secondary outcome measure 11 | 48 weeks
21. Total NSAID volume (PRISMS) in participating compared to non-participating practices | 8 weeks
22. Proportion of patients prescribed an NSAID (HIC data) stratified by age in participating compared to non-participating practices | 8 weeks
23. Proportion of patients with risk factors as defined in secondary outcome measure 1 to 9, who have been prescribed a high risk prescription as defined in outcome measure 1 to 9 and have received such a prescription within the previous 12 months | 8 weeks
24. Proportion of patients with risk factors as defined in secondary outcome measure 1 to 9, who have been prescribed a high risk prescription as defined in outcome measure 1 to 9 and have NOT received such a prescription within the previous 12 months | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Guthrie, PhD, Principal Investigator — University of Dundee
Locations (2):
- United Kingdom (2):
  - NHS Fife, General Practices Across Fife
  - NHS Tayside, General Practices Across Tayside

IPD SHARING:
Plan to Share IPD: Undecided
Follow up data is routinely collected clinical data. The trial team are data processors not data controllers, so cannot make the decision to share, although an application to share can be made to the National Health Service data controllers.

REFERENCES:
- [Background] Howard RL, Avery AJ, Slavenburg S, Royal S, Pipe G, Lucassen P, Pirmohamed M. Which drugs cause preventable admissions to hospital? A systematic review. Br J Clin Pharmacol. 2007 Feb;63(2):136-47. doi: 10.1111/j.1365-2125.2006.02698.x. Epub 2006 Jun 26. PMID 16803468
- [Background] Zullo A, Hassan C, Campo SM, Morini S. Bleeding peptic ulcer in the elderly: risk factors and prevention strategies. Drugs Aging. 2007;24(10):815-28. doi: 10.2165/00002512-200724100-00003. PMID 17896831
- [Background] Delaney JA, Opatrny L, Brophy JM, Suissa S. Drug drug interactions between antithrombotic medications and the risk of gastrointestinal bleeding. CMAJ. 2007 Aug 14;177(4):347-51. doi: 10.1503/cmaj.070186. PMID 17698822
- [Background] Hart J, Hawkey CJ, Lanas A, Naesdal J, Talley NJ, Thomson AB, Yeomans ND. Predictors of gastroduodenal erosions in patients taking low-dose aspirin. Aliment Pharmacol Ther. 2010 Jan;31(1):143-9. doi: 10.1111/j.1365-2036.2009.04133.x. PMID 19709095
- [Background] Loboz KK, Shenfield GM. Drug combinations and impaired renal function -- the 'triple whammy'. Br J Clin Pharmacol. 2005 Feb;59(2):239-43. doi: 10.1111/j.0306-5251.2004.2188.x. PMID 15676048
- [Background] Harirforoosh S, Jamali F. Renal adverse effects of nonsteroidal anti-inflammatory drugs. Expert Opin Drug Saf. 2009 Nov;8(6):669-81. doi: 10.1517/14740330903311023. PMID 19832117
- [Background] Guthrie B, McCowan C, Davey P, Simpson CR, Dreischulte T, Barnett K. High risk prescribing in primary care patients particularly vulnerable to adverse drug events: cross sectional population database analysis in Scottish general practice. BMJ. 2011 Jun 21;342:d3514. doi: 10.1136/bmj.d3514. PMID 21693525
- [Background] Avery A, Rodgers S. The PINCER trial ('A cluster randomised trial to determine the effectiveness, costs/benefits and acceptability of a pharmacist-led, IT-based intervention compared with simple feedback in reducing rates of clinically important instances of potentially hazardous prescribing and medicines management in general practice'): final report. Nottingham, University of Nottingham 2010.
- [Background] Brown CA, Lilford RJ. The stepped wedge trial design: a systematic review. BMC Med Res Methodol. 2006 Nov 8;6:54. doi: 10.1186/1471-2288-6-54. PMID 17092344
- [Derived] Grant A, Bugge C, Wells M. Designing process evaluations using case study to explore the context of complex interventions evaluated in trials. Trials. 2020 Nov 27;21(1):982. doi: 10.1186/s13063-020-04880-4. PMID 33246496
- [Derived] Dreischulte T, Grant A, Hapca A, Guthrie B. Process evaluation of the Data-driven Quality Improvement in Primary Care (DQIP) trial: quantitative examination of variation between practices in recruitment, implementation and effectiveness. BMJ Open. 2018 Jan 5;8(1):e017133. doi: 10.1136/bmjopen-2017-017133. PMID 29306877
- [Derived] Grant A, Dreischulte T, Guthrie B. Process evaluation of the Data-driven Quality Improvement in Primary Care (DQIP) trial: case study evaluation of adoption and maintenance of a complex intervention to reduce high-risk primary care prescribing. BMJ Open. 2017 Mar 10;7(3):e015281. doi: 10.1136/bmjopen-2016-015281. PMID 28283493
- [Derived] Grant A, Dreischulte T, Guthrie B. Process evaluation of the data-driven quality improvement in primary care (DQIP) trial: active and less active ingredients of a multi-component complex intervention to reduce high-risk primary care prescribing. Implement Sci. 2017 Jan 7;12(1):4. doi: 10.1186/s13012-016-0531-2. PMID 28061794
- [Derived] Dreischulte T, Donnan P, Grant A, Hapca A, McCowan C, Guthrie B. Safer Prescribing--A Trial of Education, Informatics, and Financial Incentives. N Engl J Med. 2016 Mar 17;374(11):1053-64. doi: 10.1056/NEJMsa1508955. PMID 26981935
- [Derived] Grant AM, Guthrie B, Dreischulte T. Developing a complex intervention to improve prescribing safety in primary care: mixed methods feasibility and optimisation pilot study. BMJ Open. 2014 Jan 21;4(1):e004153. doi: 10.1136/bmjopen-2013-004153. PMID 24448848
- [Derived] Grant A, Treweek S, Dreischulte T, Foy R, Guthrie B. Process evaluations for cluster-randomised trials of complex interventions: a proposed framework for design and reporting. Trials. 2013 Jan 12;14:15. doi: 10.1186/1745-6215-14-15. PMID 23311722
- [Derived] Grant A, Dreischulte T, Treweek S, Guthrie B. Study protocol of a mixed-methods evaluation of a cluster randomized trial to improve the safety of NSAID and antiplatelet prescribing: data-driven quality improvement in primary care. Trials. 2012 Aug 28;13:154. doi: 10.1186/1745-6215-13-154. PMID 22929598
- [Derived] Dreischulte T, Grant A, Donnan P, McCowan C, Davey P, Petrie D, Treweek S, Guthrie B. A cluster randomised stepped wedge trial to evaluate the effectiveness of a multifaceted information technology-based intervention in reducing high-risk prescribing of non-steroidal anti-inflammatory drugs and antiplatelets in primary medical care: the DQIP study protocol. Implement Sci. 2012 Mar 23;7:24. doi: 10.1186/1748-5908-7-24. PMID 22444945